CLINICAL TRIAL: NCT05127473
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of a Single Subcutaneous Dose of Reformulated NNC0365-3769 (Mim8) in Healthy Male Participants
Brief Title: A Research Study of How a New Medicine NNC0365-3769 (Mim8) Works in the Body of Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN7769-4882; U1111-1266-4001 (Other: World Health Organization (WHO)); 2021-003182-35 (EudraCT Number)
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers - Haemophilia A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Dose level 1 (Experimental): All participants will receive a single dose of Mim8
  Interventions: Drug: Mim8 B, 10 mg/mL; Drug: Mim8 B, placebo
- Dose level 2 (Experimental): All participants will receive a single dose of Mim8
  Interventions: Drug: Mim8 B, 10 mg/mL
- Dose level 3 (Experimental): All participants will receive a single dose of Mim8
  Interventions: Drug: Mim8 B, 100 mg/mL; Drug: Mim8 B, placebo
- Dose level 4 (Experimental): All participants will receive a single dose of Mim8
  Interventions: Drug: Mim8 B, 10 mg/mL
- Dose level 5 (Experimental): All participants will receive a single dose of Mim8
  Interventions: Drug: Mim8 B, 100 mg/mL; Drug: Mim8 B, placebo
- Dose level 6 (Experimental): All participants will receive a single dose of Mim8
  Interventions: Drug: Mim8 B, 10 mg/mL
- Dose level 7 (Experimental): All participants will receive a single dose of Mim8
  Interventions: Drug: Mim8 B, 100 mg/mL
- Dose level 8 (Experimental): All participants will receive a single dose of Mim8
  Interventions: Drug: Mim8 B, 100 mg/mL; Drug: Mim8 B, placebo
- Dose level 9 (Experimental): All participants will receive a single dose of Mim8
  Interventions: Drug: Mim8 B, 100 mg/mL; Drug: Mim8 B, placebo
- Dose level 10 (Experimental): All participants will receive a single dose of Mim8
  Interventions: Drug: Mim8 B, 100 mg/mL
- Dose level 11 (Experimental): All participants will receive a single dose of Mim8
  Interventions: Drug: Mim8 B, 100 mg/mL; Drug: Mim8 B, placebo
- Dose level 12 (Experimental): All participants will receive a single dose of Mim8
  Interventions: Drug: Mim8 B, 100 mg/mL

INTERVENTIONS:
Drug: Mim8 B, 10 mg/mL — All participants will receive a single dose of Mim8 subcutaneously (s.c- under the skin) and will stay in-house at the site until 3 days after dosing.
  Other Names: NN0365-3769
  Arms: Dose level 1; Dose level 2; Dose level 4; Dose level 6
Drug: Mim8 B, 100 mg/mL — All participants will receive a single dose of Mim8 subcutaneously (s.c- under the skin) and will stay in-house at the site until 3 days after dosing.
  Other Names: NN0365-3769
  Arms: Dose level 10; Dose level 11; Dose level 12; Dose level 3; Dose level 5; Dose level 7; Dose level 8; Dose level 9
Drug: Mim8 B, placebo — Placebo will be used to dilute the IMP to different Mim8 concentrations
  Arms: Dose level 1; Dose level 11; Dose level 3; Dose level 5; Dose level 8; Dose level 9

SUMMARY:
NN0365-3769 (Mim8) is a study medicine with the potential to prevent and reduce bleeding in people with haemophilia A (an inherited disorder in which blood does not coagulate properly).

This study will investigate if different doses of Mim8 are safe, and also check how Mim8 behaves in the body.

Twelve different doses will be tested. Participants will only get one of the doses. Which dose participants get is decided by chance. Participants will get a single injection under the skin of the belly by means of a syringe and a needle.

The study will last for about 17 - 21 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 18-55 years (both inclusive) at the time of signing informed consent
* Body mass index between 18.5 and 29.9 kg/m^2 (both inclusive)
* Body weight between 60.0 to 100.0 kg (both inclusive)
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Increased risk of thrombosis, e.g. known history of personal or first-degree relative(s) with unprovoked deep vein thrombosis
* Any clinical signs or established diagnosis of venous or arterial thromboembolic disease
* Factor VIII activity greater than or equal to150% at screening
* Any of the thrombophilia markers listed below:

  * Protein C, protein S or antithrombin below the lower normal laboratory range
  * Factor II activity, activated protein C resistance, lupus anticoagulant, anti-cardiolipin antibody (IgG and IgM) or anti-β2 glycoprotein I antibody (IgG and IgM) outside the normal laboratory range at screening

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-05-14 (Actual); Study Completion 2022-05-14 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events | From time of dosing (day 1) to day 113
  Count

SECONDARY OUTCOMES:
Number of injection site reactions | From time of dosing (day 1) to day 113
  Count
Cmax, SD: the maximum concentration of Mim8 after a single dose | From time of dosing (day 1) to day 113
  messured in μg/mL
AUC0-inf, SD: the area under the Mim8 concentration-time curve from time 0 to infinity after a single dose | From time of dosing (day 1) to day 113
  messured in μg*day/mL
t1/2, SD: the terminal half-life of Mim8 after a single dose | From time of dosing (day 1) to day 113
  messured in days
tmax, SD: the time to maximum concentration of Mim8 after a single dose | From time of dosing (day 1) to day 113
  messured in days
Change in activated partial thromboplastin time | From baseline (day 1) to day 113
  messured in seconds

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Germany (2):
  - Novo Nordisk Investigational Site, Mainz
  - Novo Nordisk Investigational Site, Neuss

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com